CLINICAL TRIAL: NCT04784338
Title: A Virtual Weight Management Shared Medical Appointment: a Feasibility Study
Brief Title: Virtual Weight Management Shared Medical Visit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided not to implement the research but instead to conduct a quality improvement project to focus on the practice of shared medical appointments (SMAs) and how to optimize them for clinical practice.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-40982
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Culinary medicine; Teaching kitchens; Virtual shared medical appointments (SMA); Mind body exercises; Social Determinants of Health (SDoH)
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual shared teaching kitchen program (Experimental): Participants will participate in virtual shared medical appointments that utilize the teaching kitchen
  Interventions: Behavioral: Virtual shared medical visit; Behavioral: Nutritional classes

INTERVENTIONS:
Behavioral: Virtual shared medical visit — a shared medical visit done by zoom in a group, 1.5 hours
Behavioral: Nutritional classes — A cooking class done by the teaching kitchen demonstrating cooking skills

SUMMARY:
Culinary medicine has emerged which provides the practical application of nutrition education through experiential learning. Studies have shown that patients with metabolic syndrome who underwent a series of classes that featured nutrition recommendations and cooking classes had weight loss, and improved cardiac health and blood sugar management.

Given the increasing focus on providing remote experiences to minimize contact and risk of infection with Sars-COV2, this pilot study at Boston Medical Center (BMC) will integrate a physician consultation, interactive didactic presentations, nutritious cooking and mind- body exercises. Patients with obesity and metabolic syndrome can attend a virtual shared medical visit series co-taught by a registered dietician and chef and an endocrinologist and weight management specialist. Data will be collected in the form of surveys, phone interviews, chart review, and home monitoring to test both the feasibility of running such an intervention virtually and to explore whether attending this one month program with weekly remote classes/visits improves vitals including weight and blood blood pressure and other small habit changes in patients.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* BMI => 30
* Must have documented measured blood pressure, weight, height in the 12 months prior to the intervention
* Enrolled in Boston Medical Center's (BMC's) Food Pantry Program

Exclusion Criteria:

* Patients with advanced dementia or uncontrolled psychiatric disease
* Uncontrolled medical illness including severe hypertension, recent acute coronary syndrome, active malignancy or other condition that would make the subject unable to complete the study procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 1 month
  Recruitment rates will be calculated by taking the number of participants enrolled over the number eligible to participate in the program
Retention of participants | 1 month
  Attendance at each of the sessions will be documented to assess retention of participants.
Facilitators for program participation | 1 month
  An investigator created questionnaire will be used to collect information about facilitators for program participation
Barriers to program participation | 1 month
  An investigator created questionnaire will be used to collect information about barriers to program participation

SECONDARY OUTCOMES:
Change in knowledge of healthy foods | baseline, 1 month
  An investigator created questionnaire will be used to collect information about knowledge of healthy foods
Change in nutritional food intake behaviours | baseline, 1 month
  An investigator created questionnaire will be used to collect information about nutritional food intake behaviours
Change in blood pressure | baseline, 1 month
  Participants will check blood pressure at home with home blood pressure cuff and record the systolic and diastolic results on home diary
Change in fasting blood glucose level | baseline, 1 month
  Participants diagnosed with diabetes will use a home glucometer to measure fasting blood glucose levels
Change in body mass index [BMI] | baseline, 1 month
  Participants will weigh themselves at home and record their weight in a study diary. The BMI will be calculated using the formula BMI= kg/m2 where kg is a person's weight in kilograms and m2 is a person's height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Ivania Rizo, MD, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No